CLINICAL TRIAL: NCT01008826
Title: Cross-Over Broccoli Sprouts Trial - Qidong
Brief Title: Cross-Over Broccoli Sprouts Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Qidong Liver Cancer Institute (Other)
Responsible Party: Principal Investigator, Thomas Kensler, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00002015; 5P01ES006052 (NIH)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: sulforaphane; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- glucoraphanin-rich broccoli extract (Experimental)
  Interventions: Dietary Supplement: broccoli sprouts extract
- sulforaphane-rich broccoli extract (Experimental)
  Interventions: Dietary Supplement: broccoli sprouts extract

INTERVENTIONS:
Dietary Supplement: broccoli sprouts extract — Glucoraphanin-rich broccoli sprouts extract: 800 micromoles daily for 7 days dissolved in 100 mL of dilute mango juice Sulforaphane-rich broccoli sprouts extract: 150 micromoles daily for 7 days dissolved in 100 mL of dilute mango juice

SUMMARY:
The study hypothesis tested is that broccoli sprouts are effective at altering the urinary levels of metabolites of the hepatocarcinogen aflatoxin B1 and of the air-borne pollutant phenanthrene in residents of Qidong, PRC, where exposures are unavoidable and high. The study will evaluate which of two formulations of broccoli sprouts beverage, glucoraphanin-rich or sulforaphane-rich, exhibits the best bioavailability and is most effective at modulating the biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25-65 in good general health with no history of a chronic illness
* normal liver function tests (ALT, AST, bilirubin)
* normal renal function tests (creatinine, BUN, urinalysis)
* serum alpha-fetoprotein negative

Exclusion Criteria:

* personal history of cancer, except for non-melanoma skin cancer
* use of prescribed medications
* hepatomegaly by clinical exam
* unwillingness to avoid cruciferous vegetable consumption for the duration of the study
* for women, a positive pregnancy test.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Urinary levels of glucoraphanin or sulforaphane and metabolites. | Endpoints will be assessed on urine samples collected daily during the intervention.

SECONDARY OUTCOMES:
Urinary levels of aflatoxin-DNA adducts and mercapturic acids as well as mercapturic acids of air-borne pollutants | Endpoints will be assessed on urine samples collected daily during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Kensler, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Qidong Liver Cancer Institute, Qidong, Jiangsu, China